CLINICAL TRIAL: NCT06060860
Title: Comparing Cognitive-Behavioral Therapy Versus Mindfulness-Based Therapy for Autistic Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Virginia (Other); Augusta University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0871
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Depression; Anxiety
Keywords: autism spectrum disorder; depression; anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT) (Active Comparator): The arm receives the Unified Protocol (UP), a modular transdiagnostic CBT treatment that uses a parsimonious approach to treatment by addressing common emotion-related mechanisms underlying both anxiety and depression.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT)
- Mindfulness-Based Cognitive Therapy (MBCT) (Active Comparator): Mindfulness-Based Cognitive Therapy (MBCT) is an empirically supported treatment that focuses on non-judgmental acceptance of present moment experiences and emotions. MBCT was adapted from Mindfulness-Based Stress Reduction (MBSR) to focus on improving mental health more specifically in individuals with depression and other psychiatric conditions.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT) — The UP incorporates common principles among empirically supported CBT protocols, including restructuring maladaptive cognitions, changing maladaptive behaviors, preventing emotion avoidance, and incorporating exposure. It consists of five core treatment modules:
  1. emotion awareness,
  2. cognitive appraisal & reappraisal,
  3. emotion avoidance & emotion-driven behaviors,
  4. awareness and tolerance of emotion-related physical sensations, &
  5. interoceptive and situational emotion-focused exposures.
  There are two introductory modules on enhancing motivation and understanding of emotional experiences. A final module is on maintenance and relapse prevention. Modules are delivered at a flexible pace and some patients may spend multiple sessions on the same module. The total number of sessions varies from patient to patient, generally ranging from 12-18 sessions (50-60 minutes) delivered weekly. All sessions are 1:1 via telehealth.
  Other Names: CBT
  Arms: Cognitive-Behavioral Therapy (CBT)
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — The study MBCT protocol is a 9-week program (90-120 minute sessions) with home-based practice between sessions. MBCT sessions incorporate formal mindfulness meditation practices such as sitting meditation, mindful movement, and body scan (with a focus on mindful and non-judgmental attention to sensations, thoughts, and feelings), as well as informal practices and homework to integrate mindful awareness into everyday life, such as mindful eating, mindful walking, and mindful breathing. All sessions are 1:1 via telehealth.
  Other Names: MBCT
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)

SUMMARY:
Autistic adults are at a greater risk for mental health problems compared to the general population, with 50% meeting criteria for a co-occurring psychiatric condition. Depression and anxiety are the most common of these conditions among autistic adults, contributing to long-term detrimental effects on health, day-to-day functioning, and quality of life. This study will conduct the first large-scale head-to-head comparison of the two most widely studied mental health interventions for autistic adults: cognitive-behavioral therapy (CBT) and mindfulness-based therapy (MBT). Both interventions are well-established, empirically supported treatments for depression and anxiety in the general population, and both interventions have demonstrated efficacy among autistic adults. However, their comparative effectiveness and heterogeneity of treatment effects have not been established in autistic adults. Both interventions will be delivered by telehealth.

DETAILED DESCRIPTION:
This study includes three aims:

Aim 1. Evaluate the effectiveness of two different mental health interventions, CBT versus MBT, to improve patient-centered mental health outcomes, quality of life, well-being, and functional impairment among autistic adults with co-occurring anxiety and/or depressive disorders.

Aim 2. Explore patient characteristics (e.g., expressive language ability, intellectual ability, alexithymia, sensory sensitivity) that may moderate the relationship between CBT or MBT and patient outcomes.

Aim 3. Compare implementation outcomes of acceptability and feasibility of CBT relative to MBT as reported by patients and clinicians using mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Co-occurring depression and/or anxiety as determined by a total score ≥10 on the PHQ-ADS
* Living in North Carolina or Virginia
* Ability to participate in therapy sessions over telehealth
* English-speaking
* Provide proof of a professional diagnosis of autism OR meet or exceed clinical cut-off on the Social Responsiveness Scale (SRS-2) autism screening instrument

Exclusion Criteria:

* Altered mental status that precludes the ability to provide informed assent or consent (acute psychosis, intoxication, or mania)
* Imminent risk of suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety and depression symptoms | Baseline, up to 18 weeks
  The Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS) is a 16-item composite measure that provides a single composite score for depression and anxiety. It comprises the 9-item Patient Health Questionnaire depression scale (PHQ-9) and the 7-item Generalized Anxiety Disorder scale (GAD-7). PHQ-ADS scores can range from 0 to 48 with higher scores indicating more severe depression/anxiety.

SECONDARY OUTCOMES:
Change in mental health | Baseline through 6 months of follow-up
  A patient-centered, single-item Participant Global Rating of Change asks participants to rate their depression/anxiety compared to how it was at the beginning of treatment on a 5-point scale (much better, a bit better, no different, a bit worse, or much worse). The score ranges from 1-5, with higher scores indicate improved depression/anxiety.
Change in psychiatric diagnosis | Baseline through 6 months of follow-up
  The Mini-International Neuropsychiatric Interview (MINI) is a widely used, structured clinical interview that was developed as a brief (~15 min), yet comprehensive, assessment of the most common psychiatric diagnoses. The MINI identifies if participants meet diagnostic criteria for major psychiatric disorders. It has 16 modules looking at 24 potential current (within the past 2 weeks or past month) and/or previous psychiatric diagnoses. Questions are rated dichotomously (yes/no) and no score is calculated. Change in total number of current psychiatric diagnoses by participant will be tracked.
Change in quality of life | Baseline through 6 months of follow-up
  The Outcome Rating Scale (ORS) is a 4-item visual analog scale assessing functioning in individual, interpersonal, social, and overall functioning over the past week. Item scores range from 0-10, with higher scores indicating better functioning.
Change in well-being | Baseline through 6 months of follow-up
  The Patient Reported Outcomes Measurement Information System (PROMIS) is a comprehensive battery of patient-centered measures. The PROMIS Autism Battery - Lifespan (PAB-L), a subset of PROMIS measures, has been validated for the assessment of autistic adults. Items are rated on either a 1 to 7 scale (5 items) or a 1-5 scale (23 items), with total scores ranging from 28 to 150, and higher scores indicating better well-being.
Change in self-acceptance | Baseline through 6 months of follow-up
  The 10-item Rosenberg Self-Esteem Scale (RSE) assesses overall self-acceptance. Item scores range from 1 to 4, with total scores ranging from 10-40, with higher scores indicating higher self-esteem.
Change in functional impairment | Baseline through 6 months of follow-up
  The brief Sheehan Disability Scale (SDS) will be used to assess the extent to which participants' mental health symptoms have disrupted their day-to-day functioning. The SDS is a 3-item discretized visual analog scale assessing functional disability in work/school, social life, and family life/home responsibilities. Scores range from 0-30, with higher scores indicating a higher degree of functional impairment.
Change in disability | Baseline through 6 months of follow-up
  The World Health Organization Disability Assessment Schedule II (WHODAS II) is a brief, 12-item measure of global disability assessing activity limitations and participation. Scores range 12 to 60, where higher scores indicate higher disability or loss of function.
Potential Negative Effects of Intervention | Up to 6-months follow-up
  The 20-item Negative Effects Questionnaire (NEQ) measures potential negative effects of psychological treatments. Scores can range from 0 to 80, with higher scores indicating more negative effects.
Intervention services satisfaction | Up to 18 weeks
  Participants will complete the Client Satisfaction Questionnaire (CSQ-8), an 8-item measure of psychotherapy satisfaction. Scores range from 8 to 32, with higher scores indicating higher satisfaction.
Intervention therapist and therapy satisfaction | Up to 18 weeks
  Participants will complete the Survey of Autism Mental Healthcare Satisfaction (SAMHS) to assess specific aspects of mental healthcare important to autistic adults. Scores range from 42-210, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Klinger, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Micah Mazurek, PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that support the results will be shared after the publication of the final research report, for a period of at least 7 years, provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of the final research report and continuing for a period of at least 7 years.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- See also: Patient-Centered Outcomes Research Institute (PCORI) Project Summary Site — https://www.pcori.org/research-results/2022/comparing-cognitive-behavioral-therapy-versus-mindfulness-based-therapy-autistic-adults